CLINICAL TRIAL: NCT03404180
Title: Peripheral Nerve Blocks for Upper Leg Amputations
Brief Title: Peripheral Nerve Blocks for Above-the-knee Amputations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201702402; OCR18952 (Other: University of Florida)
Record Dates: First submitted 2017-12-20; First posted 2018-01-19 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Vascular Diseases; Hyperglycaemia (Diabetic); Hypertension; Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Peripheral Vascular Diseases; Hyperglycemia; Hypertension; Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Pilot clinical trial with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peripheral nerve block (Experimental): Prospectively evaluate peripheral nerve blocks as a primary anesthetic in the setting of above-the-knee amputations.
  All enrollees will be administered Intravenous sedatives using propofol or dexmedetomidine and have ultrasound-guided femoral and sciatic nerve blocks placed per current practice at research site. Single-injection obturator nerve blocks and lateral femoral cutaneous nerve blocks will also be performed.
  Interventions: Procedure: Peripheral nerve block; Drug: Intravenous Sedatives; Procedure: Lateral femoral cutaneous nerve blocks; Procedure: Obturator nerve blocks

INTERVENTIONS:
Procedure: Peripheral nerve block — All enrollees will have ultrasound-guided femoral and sciatic nerve blocks placed per current practice at research site. Single-injection obturator and lateral femoral cutaneous nerve blocks will also be performed.
Drug: Intravenous Sedatives — Intravenous sedation using propofol or dexmedetomidine will be administered.
  Other Names: Propofol or Dexmedetomidine
Procedure: Lateral femoral cutaneous nerve blocks — After administration of intravenous sedation, lateral femoral cutaneous and obturator nerve blocks (in addition to the femoral and sciatic catheters) will be performed under ultrasound guidance.
Procedure: Obturator nerve blocks — After administration of intravenous sedation, lateral femoral cutaneous and obturator nerve blocks (in addition to the femoral and sciatic catheters) will be performed under ultrasound guidance.

SUMMARY:
Surgery performed with nerve blocks and sedation may be safer and provide better pain control compared to general anesthesia and opioid therapy in high-risk patient populations such as elderly and troubled with peripheral vascular disease, diabetes, hypertension, coronary artery disease, and chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Avoidance of general anesthesia in certain high-risk patient populations may have additional benefits beyond improved postoperative pain scores and analgesic consumption. The primary objective of this research will be to evaluate the ability of the femoral, sciatic, lateral femoral cutaneous nerve (LFCN), and obturator blocks to provide surgical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing above-the-knee amputation or knee disarticulation
* Ability to understand and provide informed consent

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* True allergy, not sensitivity, to any of the following substances:
* - Local anesthetics
* - Propofol or other sedative agents
* - General anesthetic agents
* Pregnancy
* Severe hepatic impairment
* Evidence of infection at or near the proposed needle insertion site
* Any sensorimotor deficit, whether acute or chronic, as determined by the PI
* Chronic use of opioid medication
* BMI ≥ 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José R Soberón, MD, Principal Investigator — Malcom Randall VA Medical Center
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peripheral Nerve Block: Prospectively evaluate peripheral nerve blocks as a primary anesthetic in the setting of above-the-knee amputations.
  All enrollees will be administered ultrasound-guided femoral and sciatic nerve placed per current practice at research site. Single-injection obturator nerve blocks and lateral femoral cutaneous nerve blocks will also be performed.
  Peripheral nerve block: All enrollees will have ultrasound-guided femoral and sciatic nerve blocks placed per current practice at research site. Single-injection obturator and lateral femoral cutaneous nerve blocks will also be performed.
  Lateral femoral cutaneous nerve blocks: After administration of intravenous sedation, lateral femoral cutaneous and obturator nerve blocks (in addition to the femoral and sciatic catheters) will be performed under ultrasound guidance.
  Obturator nerve blocks: After administration of intravenous sedation, lateral femoral cutaneous and obturator nerve blocks (in addition to the femoral and sciatic catheters) will be performed under ultrasound guidance.
Period: Overall Study
Arm/Group | Peripheral Nerve Block
Started | 30
Completed | 30 (December 18th, 2024)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peripheral Nerve Block
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Nerve Block Success as a Primary Anesthetic
Time Frame: Intraoperative period (typically one to three hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Block
Number analyzed (Participants) | 30
Participants | 1

2. Secondary Outcome: Mortality
Description: The medical record will be reviewed to assess 30-day mortality.
Time Frame: Changes from baseline through 30 days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Nerve Block
Number analyzed (Participants) | 30
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from informed consent until 30 days after surgery. Active adverse events assessments occurred at Day 30 post-enrollment (±7 days).
Arm/Group | Peripheral Nerve Block
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03404180/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT03404180/ICF_001.pdf